CLINICAL TRIAL: NCT03755492
Title: Initiative to Minimize Disparities in Postoperative Prostate Cancer Care
Status: Terminated | Type: Observational
Why Stopped: COVID related impact on recruitment. Change in treatment (more effective surgical technique ) eliminated the studied side effect, thus making the intervention arm obsolete.
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Serge Ginzburg, MD, Urologic Oncologist, Albert Einstein Healthcare Network
Other Study IDs: 5108
Record Dates: First submitted 2018-10-03; First posted 2018-11-28 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Post Prostatectomy
MeSH Terms: interventions — Absorbent Pads

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Group 1 (Provided absorbent pads): Patients will receive a 6 month supply (as needed) of absorbent pads for urinary incontinence.
  Interventions: Other: Absorbent pad for urinary incontinence
- Group 2 (not provided absorbent pads): Patients enrolled in the control arm will not receive absorbent pads.

INTERVENTIONS:
Other: Absorbent pad for urinary incontinence — 6 month supply provided to patients as needed for urinary incontinence after radical prostatectomy
  Groups: Group 1 (Provided absorbent pads)

SUMMARY:
Einstein Healthcare Network in North Philadelphia serves a predominantly underserved medical community. The investigators routinely see patients who cannot afford absorbent pads after prostate surgery, which helps with quality of life secondary to urinary incontinence. The investigators will provide absorbent pads to participants who would be unable to afford them. The investigators hypothesize that providing absorbent pads for 6 months will result in improved quality of life in regards to management of urinary incontinence after radical prostatectomy.

DETAILED DESCRIPTION:
When detected early and managed with appropriate surgical treatment, such as radical prostatectomy, Prostate cancer prognosis is excellent, but recovery may be associated with significant transient impact on quality of life. This impact most often manifests in urinary domains, specifically, development of stress urinary incontinence. Several simple, low-cost but high-yield interventions may dramatically improve patient's postoperative quality of life. However, such interventions may be out of reach for patients from Health Enterprise Zones (HEZ) with limited funds. To make resources readily available for this patient population, the inclusion criteria will be prostatectomy patients of any age who reside within the designated North Broad street HEZ.

Stress urinary incontinence after prostatectomy is a source of major distress. Incontinence tends to improve over time with most patients regaining their urinary function. Symptomatic support with disposable absorbent pads/diapers for several months helps men effectively manage this side effect. While for most men the cost of the diapers is manageable, for men in HEZ this represents a significant financial burden on the patient and on caregivers. As a result, these patients often choose to remain home bound until they recover urinary control, preventing them from early return to employment and resulting in social isolation. The Healthcare Disparity SEED Grant will provide up to a 6-month supply of disposable absorbent pads/diapers to those patients meeting our inclusion criteria. Michigan Incontinence Symptom Index (M-ISI) questionnaires will be distributed to patients pre-operatively and during interval post-operative office visits to assess patient satisfaction with voiding function.

In addition to distributing M-ISI questionnaires, we will also distribute the Extended Prostate Cancer Index Composite for Clinical Practice (EPIC-CP) to evaluate overall quality of life. This is a validated questionnaire capable of accurately assessing multiple domains of quality of life after prostate cancer treatment. Results of M-ISI and EPIC-CP scores will be compiled and analyzed to determine if intervention has resulted in measurable improvement between the treatment and control groups.

ELIGIBILITY:
Inclusion Criteria:

1. History of prostate cancer
2. Scheduled for radical prostatectomy during a designated academic year
3. Reside within Health Enterprise Zone (HEZ) of North Broad Street
4. Median annual household income < $50,000
5. Patient feels that they would struggle to afford absorbent pads and Tadalafil based on their annual income
6. Patient must have no history of stress urinary incontinence prior to surgery

Exclusion Criteria

1. Patient's who do not meet the inclusion criteria above
2. Patients who meet all inclusion criteria above, but do not want to use absorbent pads secondary to history of hypersensitivity/allergy to absorbent pads
3. Patients with cognitive impairment will be excluded from the study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Patients undergoing radical prostatectomy
Study Population: Males who reside in the health enterprise zone of north Philadelphia and are undergoing radical prostatectomy
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Michigan Incontinence Symptom Index (M-ISI) | 6 months after radical prostatectomy
  Questionnaire to assess severity of urinary incontinence and how it influences a patient's quality of life. The questionnaire asks a total of 10 questions scaled 0 to 4. The 10 questions that make up the questionnaire cover bothersome lower urinary tract symptoms specific to stress urinary incontinence, urge urinary incontinence, how many pads patients are using to manage their incontinence, and how it is influencing their daily activities. Patients with higher scores have more severe and bothersome urinary incontinence.
Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP) | 6 months after radical prostatectomy
  Questionnaire to help assess overall quality of life in patients with prostate cancer. This questionnaire is a 1-page, 16-item questionnaire that is designed to assess urinary incontinence, urinary irritation, bowel irritation, sexual health and hormonal health after prostate cancer surgery. Each domain is scored separately from a scale of 0 to 12. The minimum symptom score in each domain is a 0 and the maximum symptom score in each domain is a 12.

CONTACTS AND LOCATIONS:
Overall Officials: Serge Ginzburg, M.D., Study Director — Einstein Healthcare Network
Locations (1):
- Albert Einstein Healthcare Network, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The only time that individual participant data will be shared with other researchers is if it is requested and required by a reviewer of our research to aide with publication of our results

REFERENCES:
- [Background] Suskind AM, Dunn RL, Morgan DM, DeLancey JO, McGuire EJ, Wei JT. The Michigan Incontinence Symptom Index (M-ISI): a clinical measure for type, severity, and bother related to urinary incontinence. Neurourol Urodyn. 2014 Sep;33(7):1128-34. doi: 10.1002/nau.22468. Epub 2013 Aug 14. PMID 23945994
- [Background] Chipman JJ, Sanda MG, Dunn RL, Wei JT, Litwin MS, Crociani CM, Regan MM, Chang P; PROST-QA Consortium. Measuring and predicting prostate cancer related quality of life changes using EPIC for clinical practice. J Urol. 2014 Mar;191(3):638-45. doi: 10.1016/j.juro.2013.09.040. Epub 2013 Sep 25. PMID 24076307
- [Background] Wagner AA, Cheng PJ, Carneiro A, Dovirak O, Khosla A, Taylor KN, Crociani CM, McAnally KC, Percy A, Dewey LE, Sanda MG, Chang P. Clinical Use of Expanded Prostate Cancer Index Composite for Clinical Practice to Assess Patient Reported Prostate Cancer Quality of Life Following Robot-Assisted Radical Prostatectomy. J Urol. 2017 Jan;197(1):109-114. doi: 10.1016/j.juro.2016.07.080. Epub 2016 Jul 27. PMID 27475967